CLINICAL TRIAL: NCT02904668
Title: Effects of a Self-management Program in Patients With Chronic Neck Pain
Brief Title: Self-management Program in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0061UG
Record Dates: First submitted 2016-09-02; First posted 2016-09-19 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Neck Pain
Keywords: chronic pain
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Patients allocated to the experimental group were included in a self-management program and manual therapy program
  Interventions: Other: self-managmeent program
- Control group (Active Comparator): The intervention consisted of 45-minute manual therapy sessions. Manual therapy included "hands-on" muscular mobilization techniques (aimed at improving soft tissue function), specific articular mobilization techniques (to improve overall joint function and decrease any restrictions in movement at single or multiple segmental levels in the cervical spine), and coordination or stabilization techniques (to improve postural control, coordination, and movement patterns by using the stabilizing cervical musculature)
  Interventions: Other: self-managmeent program

INTERVENTIONS:
Other: self-managmeent program — One session was a session supervised by a physical therapist in the Faculty of Health Sciences. The program contents were educative information about chronic neck pain and healthy lifestyle habits (application of local heat/cold, and sleeping face down, using correct sitting posture, alternating body position, and using correct lifting technique (…), which were complemented by a problem-based session.

SUMMARY:
Neck pain is a complex biopsychosocial disorder often precipitated or aggravated by neck movements or sustained neck postures. The onset and course of this pain is influenced by environmental and personal factors.Many studies report that participants preferred self-care measures for the management of neck pain and they sought professional help only when those measures fail.

DETAILED DESCRIPTION:
Neck pain is the fourth leading cause of disability worldwide causing an enormous impact on individuals and their families, communities and healthcare systems.While neck pain can be severely disabling and costly, treatment options have shown moderate evidence of effectiveness. No previous study has used foam roller in patients with neck pain. In addition, it has been suggested that neurodynamic interventions provide a peripheral stimulus, reducing the pressure existing within the nerve, improving blood flow, axonal transport and nerve conduction. It was hypothesized that a self-administered intervention focused on myofascial release of main muscles related to neck pain and upper-limb active neurodynamics could reduce the presence of active trigger points and pain, improving functionality and active mobility.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain (at least 6 months' duration) not related to trauma .

Exclusion Criteria:

* Whiplash related neck pain
* Previous cervical surgical intervention
* Cognitive impairments which prevent them to follow instructions
* Visual or acoustic limitations
* Physical therapy in the previous six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Disability | Change from baseline pain at 3 weeks
  Disability will be explored using the Neck Disability Index. The patients rated their current pain and average pain over the past week on a 0-10 numerical rating scale

SECONDARY OUTCOMES:
Pain severity | Change from baseline pain at 3 weeks
  Pain will be assessed using the Brief Pain Inventory. It measures the degree of interference of pain with various aspects of life, including mobility and social activities (reactive pain) and pain severity (sensory pain).
Health related quality of life | Change from baseline health related quality of life at 4 weeks
  Health related quality of life will be measured by euroQol-5D. It contains two sections, a descriptive section and a valuation section.
Fear avoidance beliefs | Change from baseline fear avoidance beliefs at 4 weeks
  Fear avoidance beliefs will be assessed by the the Fear Avoidance Beliefs Questionnaire (FABQ). It consists of 16 sentences related to physical activity (first 5 items) and work (last 11 items).
Anxiety and depression | Change from baseline anxiety and depression at 4 weeks
  Anxiety and depression was evaluated by the the Hospital Anxiety and Depression Scale (HAD).It contains 14 items describing symptoms of depression (7 items) and anxiety (7 items)

IPD SHARING:
Plan to Share IPD: Undecided